CLINICAL TRIAL: NCT05657821
Title: THE EFFECT OF PUMPKIN SEED EXTRACT CAPSULES (Cucurbita Moschata Durch) ON NUTRITIONAL STATUS AND HAEMOGLOBIN LEVEL IN PREGNANT WOMEN TO PREVENTION STUNTING ; A PROTOCOL OF RANDOMIZED CONTROLLED TRIAL STUDY
Brief Title: The Effect Of Pumpkin Seed Extract Capsules On Nutritional Status and Haemoglobin Level in Pregnant Women.
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr. Rosdiana Syakur (Other)
Collaborators: Hasanuddin University (Other)
Responsible Party: Sponsor-Investigator, Dr. Rosdiana Syakur, Indonesia Timur University, Indonesia Timur University
Organization: Indonesia Timur University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Indonesia TimurU
Record Dates: First submitted 2022-12-11; First posted 2022-12-20 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Anemia During Pregnancy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pumpkin seed extract capsules (Experimental): . In the intervention group, pregnant women received pumpkin seed extract capsules for 12 weeks
  Interventions: Dietary Supplement: Pumpkin seeds extract capsules
- Iron tablets (Placebo Comparator): the control group received iron tablets for 12 weeks
  Interventions: Dietary Supplement: Pumpkin seeds extract capsules

INTERVENTIONS:
Dietary Supplement: Pumpkin seeds extract capsules — the intervention group was given pumpkin seed capsules for 12 weeks, and the intervention group was given iron tablets for 12 weeks

SUMMARY:
The goal of this to measure the effect of supplementation of Yellow Pumpkin Seed Extract Capsules in pregnant women on hemoglobin levels and nutritional status of pregnant women.

The main question[s] it aims to answer are:

* is there a difference in changes in nutritional status (increase in body weight and MUAC) in pregnant women who receive supplementation of Pumpkin Seed Extract Capsules and iron tablets
* is there a difference in changes in hemoglobin levels in pregnant women who receive supplementation of Pumpkin Seed Extract Capsules and iron tablets.

The research sample was divided into two groups, namely the intervention group and the control group. In the intervention group, pregnant women received pumpkin seed extract capsules for 12 weeks, while the control group received iron tablets for 12 weeks as well. Measurements of nutritional status (including measurements of body weight and Mid Upper Arm Circumference/MUAC) were carried out before and after the intervention and were monitored every month until 12 weeks when the intervention was carried out. As for measuring blood hemoglobin levels, it was taken before the intervention and after the intervention for 12 weeks

DETAILED DESCRIPTION:
This study was designed with an experimental method using a randomized double blind with a control group. The research sample was divided into two groups, namely the intervention group and the control group. In the intervention group, pregnant women received pumpkin seed extract capsules for 12 weeks, while the control group received iron tablets for 12 weeks as well. Measurements of nutritional status (including measurements of body weight and Mid Upper Arm Circumference/MUAC) were carried out before and after the intervention and were monitored every month until 12 weeks when the intervention was carried out. As for measuring blood hemoglobin levels, it was taken before the intervention and after the intervention for 12 weeks. The research will be conducted in the village of the stunting locus, Bone Regency, South Sulawesi, Indonesia. Data analysis was carried out with SPSS, where to see the difference between the intervention group and the contro group, a paired t test was used if the data was normally distributed and an alternative test if the data was not normally distributed.

ELIGIBILITY:
Inclusion Criteria:

1. in the one or second trimester of pregnancy;
2. having no complications;
3. willing to participate in this study;
4. domiciled in the stunting locus village Bone regency .

Exclusion Criteria:

* Pregnant women with complications

Ages: 17 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — pregnant woman
Enrollment: 70 (Estimated)
Dates: Start 2022-10-25 (Actual); Primary Completion 2023-01-25 (Estimated); Study Completion 2023-08-25 (Estimated)

PRIMARY OUTCOMES:
Nutritional status | 12 weeks
  measurements of body weight and Mid Upper Arm Circumference/MUAC) were carried out before and after the intervention and were monitored every month until 12 weeks when the intervention was carried out
hemoglobin levels | 12 weeks
  Hemoglobin level in the blood is measured by taking blood from the fingertip. Then measured using the digital strip method.

CONTACTS AND LOCATIONS:
Locations (1):
- Stunting Locus Village, Bone, South Sulawesi, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared with other researchers when study is done
Supporting Information: Study Protocol
Time Frame: when the study is done